CLINICAL TRIAL: NCT05322499
Title: Phase II Clinical Study of Camrelizumab Combined With Chemotherapy or Anlotinib in Second-line or Above Therapy for Advanced Esophageal Squamous Cell Cancer Previously Treated With First-line Immunotherapy
Brief Title: Phase II Clinical Study of Camrelizumab Combined With Chemotherapy or Anlotinib in Advanced Esophageal Squamous Cell Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Yu Xinmin, Physician, Zhejiang Cancer Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2021-444
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Stage IV Esophagus Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — camrelizumab; Irinotecan; Paclitaxel; Docetaxel; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined chemotherapy group (Experimental): Camrelizumab: Subjects were infused at a dose of 200 mg/time, D1, once every 3 weeks (q3w);
  Chemotherapy (considered by investigator on a patient-by-patient basis):
  Irinotecan: 100-125mg/m2, d1, d8; q21d; Paclitaxel: 135-175mg/m2, d1, Q3W; Docetaxel: 60-75mg/m2, d1, Q3W Albumin paclitaxel: 100-135mg/m2, d1, d8, Q3W. Treat until disease progression or intolerable toxicity
  Interventions: Drug: Camrelizumab; Drug: Irinotecan; Drug: Paclitaxel; Drug: Paclitaxel-albumin; Drug: Docetaxel
- Combined anlotinib group (Experimental): Camrelizumab: Subjects were infused at a dose of 200 mg/time, D1, once every 3 weeks (q3w); Anlotinib: 12mg, qd, d1-d14, q3w; Treat until disease progression or intolerable toxicity.
  Interventions: Drug: Camrelizumab; Drug: Anlotinib

INTERVENTIONS:
Drug: Camrelizumab — 200mg/dose intravenous infusion, D1, once every 3 weeks (q3w);
  Other Names: SHR-1210
Drug: Irinotecan — 100-125mg/m2，d1，d8；q21d
  Arms: Combined chemotherapy group
Drug: Paclitaxel — 135-175mg/m2，d1，Q3W
  Arms: Combined chemotherapy group
Drug: Paclitaxel-albumin — 100-135mg/m2, d1、d8，Q3W
  Arms: Combined chemotherapy group
Drug: Docetaxel — 60-75mg/m2，d1，Q3W
  Arms: Combined chemotherapy group
Drug: Anlotinib — 12mg，qd，d1-d14，q3w
  Arms: Combined anlotinib group

SUMMARY:
To observe and evaluate the efficacy and safety of camrelizumab combined with chemotherapy or anlotinib in patients with advanced esophageal squamous cell carcinoma previously Treated With First-line Immunotherapy

DETAILED DESCRIPTION:
How to improve the efficacy of immunotherapy, evaluate the results of immunotherapy more objectively, and overcome immune resistance through reasonable combined treatment methods, so as to maximize the benefit of patients from immunotherapy, is an urgent research direction to be explored. Therefore, this study intends to observe and evaluate the efficacy and safety of camrelizumab combined with chemotherapy or anlotinib in patients with advanced esophageal squamous cell cancer previously Treated With First-line Immunotherapy . It can provide a basis for the treatment of esophageal cancer after immune resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, male or female;
2. Participants signed and dated written informed consent. (Informed consent forms must be signed prior to any protocol-related procedures that are not part of the participant's routine medical care.);
3. Patients with advanced esophageal squamous cell carcinoma diagnosed as stage IV by histopathology or cytology;
4. ECOG PS score of physical condition: 0-1 points;
5. Expected survival period ≥ 3 months;
6. Patients with esophageal squamous cell carcinoma who have received first-line or above systemic therapy in the past, and who have received at least 2 times of PD-1 immunotherapy;
7. Laboratory inspection indicators meet the following requirements:

(1) Bone marrow function: hemoglobin (Hb) ≥ 90g/L; white blood cell count (WBC) ≥ lower limit of normal; absolute neutrophil value (ANC) ≥ 1.5×10^9 /L; platelet count ≥ 100×10^9 / L; (2) Renal function: Cr≤UNL (upper limit of normal)×1.5, endogenous creatinine clearance rate (Ccr)≥55 ml/min; (3) Liver function: total bilirubin≤ULN×1.5; ALT and AST≤ULN×2.5; (4) Coagulation function: the international normalized ratio of prothrombin time is less than or equal to ULN×1.5, and the partial thromboplastin time is within the normal range; 8. Females of childbearing age agree to contraception during the study period and within 6 months after the end of the study; serum or urine pregnancy test is negative within 7 days before the study is enrolled, and non-lactating patients; males agree to use contraception during the study period and within 6 months after the end of the study contraceptive patients; 9. Those who have not participated in clinical trials of other drugs within 4 weeks before enrollment; 10. Patients with good compliance are expected to be able to follow up the efficacy and adverse reactions according to the requirements of the program; 11. In view of the unclear definition of primary drug resistance and the lack of standard treatment options for such patients, there is a potential possibility of benefiting such patients with immunization combined with anti-angiogenesis or chemotherapy, but there is also a certain risk of hyperprogression; Therefore, for patients with possible primary drug resistance, they must be included in the group after evaluation by the investigator.

Exclusion Criteria:

1. Other malignant tumors have been diagnosed in the past 5 years;
2. Patients with active bleeding within two months of the primary tumor;
3. Patients with severe adverse reactions related to immunotherapy after previous use of immunotherapy;
4. Patients with any active autoimmune disease or autoimmune disease (including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, enteritis, multiple sclerosis, vascular inflammation, glomerulonephritis, uveitis, hypophysitis, hyperthyroidism, etc.). Type 1 diabetes mellitus receiving stable doses of insulin, hypothyroidism receiving only hormone replacement therapy, no systemic therapy required, and no acute exacerbation of skin disease (eg, eczema, vitiligo, or psoriasis) within 1 year prior to the screening period. );
5. Suffering from uncontrolled clinical symptoms or diseases of the heart;
6. Active infection or fever (except for definite tumor fever);
7. History or evidence of interstitial lung disease or active non-infectious pneumonia;
8. Females of childbearing age agree to contraception during the study period and within 6 months after the end of the study; serum or urine pregnancy test is negative within 7 days before the study is enrolled, and non-lactating patients; males agree to use contraception during the study period and within 6 months after the end of the study contraceptive patients;
9. Those who have not participated in clinical trials of other drugs within 4 weeks before enrollment;
10. Patients with good compliance are expected to be able to follow up the efficacy and adverse reactions according to the requirements of the program;
11. In view of the unclear definition of primary drug resistance and the lack of standard treatment options for such patients, there is a potential possibility of benefiting such patients with immunization combined with anti-angiogenesis or chemotherapy, but there is also a certain risk of hyperprogression; Therefore, for patients with possible primary drug resistance, they must be included in the group after evaluation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2023-04-15 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 24 month
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1

SECONDARY OUTCOMES:
Duration of response (DoR) | Up to 24 month
  DOR is defined as the time from first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first.
Disease control rate (DCR) | Up to 24 month
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or stable disease (SD) per RECIST 1.1.
Progression-free survival (PFS) | Up to 24 month
  Progression-free survival is defined as the duration from date of enrollment to the first occurrence of progression of disease or death from any cause
Overall survival (OS) | Up to 24 month
  Overall survival is defined as the duration from date of enrollment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Xinmin Yu, Doctor, Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No